CLINICAL TRIAL: NCT01187940
Title: Evaluating Psychoeducation for People With Autism Spectrum Disorder
Brief Title: Evaluating PEGASUS - a Group Intervention for Young People With an Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Child Health (Other)
Responsible Party: Research Governance Co-ordinator, Institute of Child Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09BS22
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Efficacy of PEGASUS
Keywords: Autism Spectrum Disorder;; Psychoeducation
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEGASUS (Experimental): PEGASUS - a psychoeducational group intervention with parallel parent and child sessions.
  Interventions: Behavioral: PEGASUS
- Placebo (No Intervention): Will receive managment as usual from their local educational and NHS services

INTERVENTIONS:
Behavioral: PEGASUS — PEGASUS - a psychoeducational group intervention with parallel parent and child sessions.
  Arms: PEGASUS

SUMMARY:
When a clinician gives an autism spectrum disorder (ASD) diagnosis they hope this will be helpful to the person receiving it and their family. In reality children with an ASD describe few benefits to receiving this diagnosis - they often report feeling confused and stigmatised by it. Parents can also struggle to understand their child's diagnosis and report needing greater support from professionals in this respect (Midence & O'neill, 1999; Osborne & Reed, 2008).

Little is known about how to help children and families integrate their ASC 'label' in a positive way. Whilst there is anecdotal evidence that psychoeducation after diagnosis can help, there has been no formal evaluation of this approach and no evidence-based programmes of this type are available. In the current study the investigators aim to test empirically a psychoeducational programme for children with an ASD ('PEGASUS'), using a randomised controlled design. The investigators aim to evaluate whether this psychological and educational intervention impacts positively upon understanding of ASC, self-esteem, functional adaption, well-being and family functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Received an ASD diagnosis from Child and Adolescent Psychiatrist, Clinical Psychologist or Paediatrician.
2. Aware of ASD diagnosis.
3. Aged between 9 and 14 years.
4. Able to function in group setting, as evidenced in educational context.
5. Speaks English

Exclusion Criteria:

1. No generalised Intellectual Disability as indicated by IQ below 65.
2. Not engaged in additional formal psychosocial intervention during study period.
3. Not taking psychiatric medication at baseline assessment, or taking a stable dose of psychiatric medication expected to remain constant throughout study participation.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Autism Knowledge Questionnaire | 30 months
  All measures taken at baseline, termination of treatment and six months follow-up.
Child Behaviour Checklist | 30 months
  All measures taken at baseline, termination of treatment and six months follow-up.
Vineland-II, Rosenburg Self-Esteem Scale | 30 months
  All measures taken at baseline, termination of treatment and six months follow-up.
Parenting Stress index | 30 months
  All measures taken at baseline, termination of treatment and six months follow-up.

SECONDARY OUTCOMES:
Qualitative interview conducted at baseline and termination. | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: William Mandy, Dr, Study Director — Institute of Child Health; David Skuse, Professor, Principal Investigator — Institute of Child Health
Locations (1):
- Institute of Child Health, London, United Kingdom

REFERENCES:
- [Derived] Gordon K, Murin M, Baykaner O, Roughan L, Livermore-Hardy V, Skuse D, Mandy W. A randomised controlled trial of PEGASUS, a psychoeducational programme for young people with high-functioning autism spectrum disorder. J Child Psychol Psychiatry. 2015 Apr;56(4):468-76. doi: 10.1111/jcpp.12304. Epub 2014 Aug 1. PMID 25132516